CLINICAL TRIAL: NCT06468579
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅰ Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics of GT20029 Gel and Solution for Single and Multi Dose External Administration in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability and PK of GT20029 Gel and Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT20029-CN-1001
Record Dates: First submitted 2024-05-27; First posted 2024-06-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-05

CONDITIONS: Acne; Alopecia
MeSH Terms: conditions — Acne Vulgaris; Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: GT20029 (Experimental)
  Interventions: Drug: GT20029
- Placebo Comparator: GT20029 Placebo (Placebo Comparator)
  Interventions: Drug: GT20029 matching placebo

INTERVENTIONS:
Drug: GT20029 — Stage 1: GT20029 gel single ascending dose (1mg, 2mg, 5mg, 10mg) with 14 days washout window; Multi ascending dose (2mg QD, 2mg Q12h, 5mg QD, 5mg Q12h,10mg QD) for 14 consecutive days; Stage 2: GT20029 solution multi ascending dose (5mg QD, 10mg QD, 20mg QD) for 14 consecutive days;
  Arms: Experimental: GT20029
Drug: GT20029 matching placebo — Stage 1: GT20029 gel matching placebo single ascending dose (1mg, 2mg, 5mg, 10mg) with 14 days washout window; Multi ascending dose (2mg QD, 2mg Q12h, 5mg QD, 5mg Q12h,10mg QD) for 14 consecutive days; Stage 2: GT20029 solution matching placebo multi ascending dose (5mg QD, 10mg QD, 20mg QD) for 14 consecutive days;
  Arms: Placebo Comparator: GT20029 Placebo

SUMMARY:
The study is a randomized, double-blind, vehicle-controlled, parallel group, phase 1 study to evaluate the Safety, Tolerability and PK of GT20029 in healthy subjects

DETAILED DESCRIPTION:
GT20029 is a new investigational androgen receptor (AR) degrader for the treatment of acne and androgenetic alopecia.

A total of 92 healthy subjects planned to be enrolled. It is divided into a single dose dosage stage and a multi dose dosage stage.

This study comprised two stages. Stage 1 included single ascending dose (SAD) and multiple ascending dose (MAD) parts. In the SAD part, 28 subjects were first enrolled to evaluate GT20029 gel or the corresponding vehicle (placebo) at four dosing levels: 1 mg, 2 mg, 5 mg, and 10 mg. In the MAD part, 40 subjects were enrolled with five dosing levels: 2 mg QD, 2 mg Q12h, 5 mg QD, 5 mg Q12h, and 10 mg QD for 14 consecutive days. SAD subjects could transfer to the MAD QD dosing cohort at the same dosing level after a 14-day wash-out period if safety was confirmed by the investigator.

In Stage 2, 24 subjects were enrolled to evaluate GT20029 solution or the corresponding vehicle (placebo) in the MAD part for 14 days with three dosing levels: 5 mg QD, 10 mg QD, and 20 mg QD. The administration site was an 8 cm by 8 cm area selected on the subjects' backs.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria may be included in this study:

1. Subjects aged 18 to 60 years (including the boundary value), male or female;
2. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 26 kg/m2 inclusive;
3. The subject voluntarily participates in the clinical trial and signs the informed consent form, is able to communicate well with the investigator, and understands and complies with the requirements of this study;
4. From signing the informed consent form to 3 months after the last dose, fertile female subjects or partners of fertile male subjects agree to and can take effective contraceptive measures, such as avoiding sex or using condoms, intrauterine device and other reliable contraceptive measures;
5. Willing to use the investigational drug as required during the trial and refrain from using any other medication while receiving the investigational drug.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Previous allergy to the investigational drug and/or any excipients, or allergic constitution (such as two or more drugs, food or pollen allergy);
2. Currently suffering from skin diseases requiring treatment and researchers believe that it is not suitable for enrollment, such as solar dermatitis, psoriasis, seborrheic dermatitis, rosacea, folliculitis, eczema and very severe acne;
3. Previous or current suffering from the following diseases and researchers believe that cannot be enrolled, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bone and other system diseases and malignant tumors;
4. Screening physical examination, vital signs, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, etc.), 12-lead ECG results are abnormal and clinically significant, and have an impact on the evaluation of this trial;
5. Subjects who plan to use various skin care products simultaneously on the back skin during the trial;
6. Blood collection difficulties or cannot tolerate venipuncture, have a history of fainting needle halo blood;
7. Blood donation or blood loss ≥ 200 mL within 3 months before screening, or plan to donate blood or blood components during the study or within 3 months after the end of the study;
8. Smoking more than 5 cigarettes per day within 3 months before screening and those who cannot abstain from smoking throughout the trial;
9. Drink more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL beer or 45 mL of spirits with 40% alcohol content or 150 mL wine) within 3 months before signing the informed consent form, or have a positive breath alcohol test on the day before administration (breath alcohol content > 0.0 mg/100 mL), or cannot abstain from alcohol during the trial;
10. Patients who have been drinking excessive tea, coffee or caffeine-containing beverages for a long time (more than 8 cups a day, 1 cup = 200 mL);
11. Consumption of any food or beverage containing caffeine, alcohol, xanthine or grapefruit ingredients (such as coffee, strong tea, chocolate, etc.) within 48 hours before the first dose;
12. Use of any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.) or health products within 14 days or 7 half-lives (whichever is the longest) before the first dose;
13. Use of any known liver enzyme inducer or liver enzyme inhibitor within 30 days before the first dose ;
14. Use of drugs with the same target and mechanism (androgen receptor degraders) within 1 month before screening;
15. Drug addiction and drug abuse test one or more positive, 1 year before the test drug abuse/dependence history or drug history;
16. Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C virus antibody, treponema pallidum antibody test positive;
17. Pregnant or lactating women or female subjects with positive blood pregnancy during screening period;
18. Subjects with back application site skin damage or wounds, tattoos or scars;
19. Planned to participate in strenuous exercise during the trial, including body contact exercise or collision exercise;
20. Major surgery within 3 months before screening, or plan to undergo major surgery during the trial;
21. Participating or participating in any drug or medical device clinical trial within 3 months before screening;
22. Unable to communicate or cooperate with medical staff due to neurological, psychiatric or language disorders;
23. Other conditions that the investigator considers unsuitable for participating in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of GT20029 for single dose and multi dose topical administration in healthy subjects. | 14 days
  Incidence of Treatment Emergent Adverse Events, as assessed by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, V2.1

SECONDARY OUTCOMES:
To characterize the peak concentration (Cmax) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, Cmax
To characterize the time to peak concentration (Tmax) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, Tmax
To characterize the elimination half-life (t1/2) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, t1/2
To characterize the area under the concentration-time curve from time zero to the last measurable concentration (AUC0-t) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, AUC0-t
To characterize the area under the concentration-time curve from time zero to infinity (AUC0-∞) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, AUC0-∞
To characterize the area under the terminal elimination rate constant (λz) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, λz
To characterize the area under the apparent volume of distribution (Vd/F) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, Vd/F
To characterize the area under the apparent clearance (CL/F) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration is: Stage 1, single-dose administration, CL/F
To characterize the area under the concentration-time curve at steady state (AUCss) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1, multi-ascending dose and Stage 2, AUCss
To characterize the peak concentration at steady state (Cmax,ss) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1, multi-ascending dose and Stage 2, Cmax,ss
To characterize the trough concentration at steady state (Cmin,ss) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1, multi-ascending dose and Stage 2, Cmin,ss
To characterize the time to peak concentration at steady state (Tmax,ss) of GT20029 | 14 days
  The plasma concentration time data for GT20029 and its metabolite will be analyzed using noncompartmental methods. Actual dosing and sampling times will be used for analyses. The primary PK parameters of interest following dose administration are: Stage 1, multi-ascending dose and Stage 2, Tmax,ss
Evaluate the ratio of systemic exposure between the gel and solution formulation. | 14 days
  Evaluate the ratio of systemic exposure between the gel and solution formulation by using GT20029 gel as a reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Research Center, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No